CLINICAL TRIAL: NCT07403396
Title: Quantitative Assessment of Static Balance in Children With Autism Spectrum Disorder Using VRRS
Brief Title: Static Balance Assessment in Children With ASD Using VRRS
Status: Recruiting | Type: Observational
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Collaborators: Messina, Italy (Other)
Responsible Party: Principal Investigator, Flavia Marino, Head of Unit, Istituto per la Ricerca e l'Innovazione Biomedica
Other Study IDs: CNR-IRIB-PRO-2026-001
Record Dates: First submitted 2026-01-13; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: Autism; Virtual Reality; Virtual Reality Rehabilitation System; Postural control
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with autism spectrum condition: Fifty ASD children aged 6 to 13 years, IQ > 60, in the absence of motor deficits due to another clinical condition.
  Interventions: Other: Virtual Reality Rehabilitation System (VRRS) in conjunction with a stabilometric balance platform

INTERVENTIONS:
Other: Virtual Reality Rehabilitation System (VRRS) in conjunction with a stabilometric balance platform — In a single session to evaluate postural control children with ASD will participate in an activity utilizing the Virtual Reality Rehabilitation System (VRRS) in conjunction with a stabilometric balance platform. During the assessment task, participants will stand on the balance platform with their eyes open, focusing on a fixed point displayed on the VRRS screen for a duration of one minute. This process will be repeated three times for each participant. The combined use of VRRS and the stabilometric balance platform aims to provide a comprehensive evaluation of postural control abilities.

SUMMARY:
Children with autism spectrum disorder (ASD) often exhibit postural and balance difficulties, which can impact daily functioning and motor development. Quantitative assessment using Virtual Reality Rehabilitation System (VRRS) provides precise measurements to better understand these deficits and their potential relationship with cognitive functioning. This observational trial aims to evaluate static balance in children with ASD aged 6-10 years. A total of 50 participants were enrolled, with 10 children in each age group. Static balance was assessed using the VRRS and a specific balance task, measuring 13 quantitative parameters including Mean Distance Centre of Pressure (MD_COP), Root Mean Square of Distance (RMS), Total Excursion (ESC), Velocity (VEL) , and Sway area (SWAY). Cognitive functioning was also recorded using standardized IQ assessments to explore correlations between balance performance and cognitive abilities. All data were stored in a dedicated database for analysis.

Participant recruitment: Children diagnosed with ASD will be recruited from the clinical facilities of the Institute for Biomedical Research and Innovation of the National Research Council of Italy (IRIB-CNR) in Messina as part of an ongoing research program.

Withdrawn criteria: Participants will be considered withdrawn if any of the following occurs: (1) participant chooses to withdraw from the study at any time, (2) intolerable adverse effects, (3) major violation of the study protocol, and (4) other circumstances that would endanger the health of the subject if he/she would to continue his/her participation in the trial.

Virtual Reality Rehabilitation system: The VRRS, a sophisticated technological innovation, aims to generate immersive and interactive settings intended for therapeutic and evaluative objectives. Through the utilization of virtual reality (VR) technology, it constructs diverse scenarios, tasks, and activities in a controlled digital environment, fostering engagement. Primarily crafted for rehabilitation purposes, the VRRS features adaptable programs addressing various therapeutic requirements, encompassing motor skill enhancement, cognitive challenges, and assessments related to balance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autism;
* QI ≥ 60

Exclusion Criteria:

* Motor deficits due to another clinical condition

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Fifty children with ASD. The children with ASD will be recruited and tested at the clinical facilities of the Institute for Biomedical Research and Innovation of the National Research Council of Italy (IRIB-CNR) in Messina. To be included in the study the child needs to have an ASD diagnosis based on the DSM-5 criteria from a licensed clinical child neuropsychiatrist but no established intellectual disability diagnosis.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01-02 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Centre of Pressure (COP) displacement | The test needs approximately 3 minutes per child
  The Virtual Reality Rehabilitation system (VRRS; Khymeia, Italy) is an innovative system based on the concept of augmented feedback. It consists of devices for clinical use and a tablet for home-based telerehabilitation, which can be remotely managed. Different peripherals can be connected via USB to the VRRS, including a stabilometric balance platform. It is a force plate (80 ×55 cm) able to detect forces in the z-direction and the Centre of Pressure (COP) displacement in millimeter (mm). The COP displacement is the distance and direction that COP moves from a reference point or position, in the anterior-posterior (AP) and medial-lateral (ML) direction, thanks to the four load cells integrated into the balance platform. Moreover, a dedicated software can be used to calibrate the balance platform which will allow the estimation of static postural data. After each measurement, a report containing a summary of the data can be exported through the dedicated software.
Centre of Pressure (COP) velocity | The test needs approximately 3 minutes per child
  The Virtual Reality Rehabilitation system (VRRS; Khymeia, Italy) is an innovative system based on the concept of augmented feedback. It consists of devices for clinical use and a tablet for home-based telerehabilitation, which can be remotely managed. Different peripherals can be connected via USB to the VRRS, including a stabilometric balance platform. It is a force plate (80 ×55 cm) able to detect Centre of Pressure (COP) velocity in millimeter per second (mm/s), a sensitive measure to detect changes in postural control.
Centre of Pressure (COP) sway area | The test needs approximately 3 minutes per child
  The Virtual Reality Rehabilitation system (VRRS; Khymeia, Italy) is an innovative system based on the concept of augmented feedback. It consists of devices for clinical use and a tablet for home-based telerehabilitation, which can be remotely managed. Different peripherals can be connected via USB to the VRRS, including a stabilometric balance platform. It is a force plate (80 ×55 cm) able to detect the Centre of Pressure (COP) sway area in square millimeter per second (mm2 /s). Sway area is the area enclosed by the COP trajectory per unit time.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Marino, Principal Investigator — Italy Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR) Messina, Italy, 98164
Locations (1):
- Italy Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR), Messina, Italy

IPD SHARING:
Plan to Share IPD: No